CLINICAL TRIAL: NCT04477057
Title: A Phase 1, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Single and Multiple Doses of Oral Administration of HS-10241 in Patients With Locally Advanced or Metastatic Solid Tumors Who Have Progressed Following Prior Therapy
Brief Title: PhaseⅠStudy of the HS-10241 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10241-101-CN
Record Dates: First submitted 2020-04-27; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor
Keywords: phase 1, solid tumor, inhibitor of c-Met kinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm (Other): one arm
  Interventions: Drug: HS-10241

INTERVENTIONS:
Drug: HS-10241 — HS-10241 is a tablet in the form of 100 mg, oral, once daily.

SUMMARY:
HS-10241 is a highly potent and selective small molecule inhibitor of c-Met kinase. In preclinical studies, it demonstrated strong activity against c-Met kinase in vitro and in vivo, and inhibited tumor cell growth. This study is conducted to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HS-10241 at single dose and multiple doses.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter study to evaluate safety, tolerability, pharmacokinetics, and efficacy of single and multiple doses of oral administration of HS-10241 in patients with locally advanced or metastatic solid tumors who have progressed following prior therapy. There is a dose-escalation study, which is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and repeat doses of HS-10241 given once every day (QD). An alternative dosing schedule of twice every day (BID) may be investigated if the drug clearance of HS-10241 is faster than anticipated.

All patients will be carefully followed for adverse events during the study treatment and for 28 days after the last dose of study drug. Subjects of this study will be permitted to continue therapy with assessments for progression once every 6 weeks, if the product is well tolerated and the subject has stable disease or better. As the disease progresses, survival follow-up is recommended bimonthly.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Men or women aged more than or equal to (≥) 18 years, and less than (<) 75 years.
3. Histologically or cytologically confirmed solid tumor, either refractory to standard therapy or for which no effective standard therapy is available.
4. ECOG performance status of 0-1, estimated life expectancy greater than (>) three months.
5. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements.
6. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening:

   1. Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory.
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
7. Male patients should be willing to use barrier contraception (i.e., condoms).

Exclusion Criteria:

1. Treatment with any of the following:

   1. Any cytotoxic chemotherapy, investigational agents, or anticancer drugs for the treatment of advanced solid tumor used for a previous treatment regimen or clinical study within 14 days of the first dose of study drug.
   2. Drugs with immunoregulatory indications within 7 days of the first dose of study drug.
   3. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
   4. Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) , unrecovered wound, ulcer, or fracture within 4 weeks of the first dose of study drug.
   5. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
   6. Previous or current treatment with drugs targeting the c-MET/HGF pathway.
2. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia.
3. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment. Meningeal or brainstem metastases.
4. Pleural or peritoneal effusion requiring clinical intervention (except for effusion stable at least 1 week after clinical intervention). Pericardial effusion (except for non-tumorous micro pericardial effusions).
5. The tumor compresses or invades important surrounding organs (such as trachea, esophagus, superior vena cava, heart, and aorta, etc), or causes significant mediastinal displacement.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the investigator's opinion, makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol such as active infection (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]). Screening for chronic conditions is not required.
7. Any active infection requiring treatment or systemic anti-infective agent used in one week prior to first dose administration.
8. Active hemoptysis, active diverticulitis, peritoneal abscess, gastrointestinal obstruction that requires clinical intervention.
9. Medical history of arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, within 6 months prior to screening. Medical history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism within 3 months prior to screening.
10. Varices of the esophagus or stomach that require immediate intervention (e.g., sclerotherapy).
11. Any life-threatening bleeding events or Grade 3 or 4 gastrointestinal/varicose bleeding events requiring blood transfusion, endoscopy, or surgical treatment occurred within 3 months prior to enrollment.
12. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.
13. Any of the following cardiac criteria:

    1. Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
    2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
    4. Left ventricular ejection fraction (LVEF) ≤ 40%.
    5. Any newly diagnosed clinically important arrhythmia which is no reasonable reason other than tumor to explain within 3 months prior to enrollment.
14. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
15. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count (ANC) <1.5×109 / L
    2. Platelet count <100×109 / L
    3. Hemoglobin <90 g/L（<9 g/dL）
    4. Alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
    5. Aspartate aminotransferase (AST) > 2.5 × ULN if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases.
    6. Total bilirubin (TBL) > 1.5 × ULN if no liver metastases or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
    7. Serum albumin (ALB) < 28 g/L, patients corrected by supplementation with human albumin should to exclude.
    8. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
    9. Urine protein ≥ 2+. When the Urine protein ≥ 2+ at baseline, 24-hour urine for collection, if the protein content in urine is less than 1g for 24 hours, inclusion is allowed.
16. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of HS-10241.
17. History of hypersensitivity to any active or inactive ingredient of HS-10241 or to drugs with a similar chemical structure or class to HS-10241.
18. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
19. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.
20. History of other primary malignancies, excluding:

    1. Malignancies that have been recovered, have been inactive for ≥5 years prior to inclusion and have a very low risk of recurrence.
    2. Non-melanoma skin cancer or malignant freckle mole with adequate treatment and no evidence of disease recurrence.
    3. Carcinoma in situ with adequate treatment and no evidence of disease recurrence.
21. Women who are breastfeeding or have a positive serum pregnancy test at Screening.
22. Any uncontrolled metabolic dysfunction, local or systemic disease that is not caused by a malignant tumor, disease or symptoms secondary to the tumor, can lead to higher medical risk and/or uncertainty in the evaluation of survival.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with any dose limiting toxicity (DLT) | From the single dose to the last dose of the first cycle defined as 21 days of multiple dosing (4 weeks).
  DLT is defined as one of the following HS-10241 related adverse event (AE) that occurs during the DLT period, excluding AE assessed by investigator exclusively related to subject's underlying disease or medical condition (graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0): Grade 4 hematological toxicity and Grade ≥ 3 non-hematological toxicity.
To determine the maximum tolerated dose (MTD) | From the single dose to the last dose of the first cycle defined as 21 days of multiple dosing (4 weeks).
  MTD was defined as the previous dose level at which 2 out of 3 subjects or 2 out of 6 subjects experienced a DLT.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, RECIST1.1, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  In the study of single-dose, Cmax will be obtained following administration of a single oral dose of HS-10241 on Day 1 to Day 6.
Observed maximum plasma concentration (Cmax ss) after multiple dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of dosing in the second 21-Day cycle of therapy
  At multiple-dose, Cmax ss will be obtained on Day 1 of dosing in the second 21-Day cycle of therapy.
Time to reach maximum plasma concentration (Tmax) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  In the study of single-dose, Tmax will be obtained following administration of a single oral dose of HS-10241 on Day 1 to Day 6.
Time to reach maximum plasma concentration (Tmax) after multiple dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1 of dosing in the second 21-Day cycle of therapy
  At multiple-dose, Tmax will be obtained on Day 1 of dosing in the second 21-Day cycle of therapy.
Apparent terminal half-life (t1/2) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to the 24 hour sampling time (AUC0-24) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  Area under the plasma concentration versus time curve from time zero to the 24 hour sampling time 24 at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-24 was to be calculated according to the mixed log-linear trapezoidal rule.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-10241 | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24,48, 72,120 hours post-dose on Day 1 single dose
  AUC0-∞ was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
To further evaluation of the anti-tumor activity of HS-10241 by assessment of objective response rate (ORR) | 0-360day
  Anti-tumoral efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors at baseline (Day -28 to -1). For patients that continue on repeat 21-Day cycles after the primary evaluation period, progression will be assessed after each 6 weeks of therapy. ORR is defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.
Duration of response of HS-10241 | 0-360day
  Duration of response assessed by RECIST 1.1. Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of a objective disease progression (PD) or death.
Time to objective response of HS-10241 | 0-360day
  Objective response was assessed by RECIST 1.1.
Disease control rate of HS-10241 | 0-360day
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmd CR, PR, or stable disease for at least 5 weeks).
Deepness of response of HS-10241 | 0-360day
  Objective response was assessed by RECIST 1.1 thereby to evaluate deepness of response. Depth of response was defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of new lesions, or progression of non-target lesions compared with baseline.
Progression-free survival of HS-10241 | 0-360day
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documention of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Principal Investigator — Shanghai Chest Hospital; Shenglin Ma, Principal Investigator — First People's Hospital of Hangzhou; Deguang Mu, Principal Investigator — Zhejiang Provincial People's Hospital; Jianhua Chen, Principal Investigator — Hunan Cancer Hospital; Xiaorong Dong, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Xiaoju Zhang, Principal Investigator — Henan Provincial People's Hospital; Xingya Li, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; 7Yubiao Guo, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No